CLINICAL TRIAL: NCT02896595
Title: General Anesthesia With Endotracheal Tube Versus Laryngeal Mask Airway in Patients Undergoing Catheter Ablation for Atrial Fibrillation, a Non-inferiority Trial
Brief Title: General Anesthesia With ETT vs LMA in Patients Undergoing Ablation for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HM20007902
Record Dates: First submitted 2016-08-29; First posted 2016-09-12 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anesthesia, General; Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Anesthesia with endotracheal tube (Active Comparator): Patients assigned to the ETT tube group will have ETT placed in the safest manner deemed appropriate by attending anesthesiologist. Possible ways to have ETT placed will be using direct laryngoscopy, glidescope or fiberoptic intubations. Size of ETT will be decided based on patient characteristics and discretion of attending anesthesiologist. Once placed, auscultation and capnography will be used to ensure correct placement of ETT.
  Interventions: Device: General Anesthesia with endotracheal tube
- General Anesthesia with laryngeal mask airway (Active Comparator): Patients assigned to the LMA group will have LMA placed in a standard fashion by anesthesia provider. LMA size will be decided based on patient characteristics and at the discretion of attending anesthesiologist. LMA used will be LMA Supreme (Teleflex Medicals, Ireland). Once placed auscultation will be used to ensure correct placement of LMA.
  Interventions: Device: General Anesthesia with laryngeal mask airway

INTERVENTIONS:
Device: General Anesthesia with endotracheal tube — Patient randomized to this arm will have general anesthesia with endotracheal tube placed and will be kept at an appropriate depth of anesthesia for patient comfort and procedure needs.
  Arms: General Anesthesia with endotracheal tube
Device: General Anesthesia with laryngeal mask airway — Patients randomized to this arm will have general anesthesia with laryngeal mask airway placed and will be kept at an appropriate depth of anesthesia for patient comfort and procedure needs.
  Arms: General Anesthesia with laryngeal mask airway

SUMMARY:
In recent years it has been shown that catheter ablation of symptomatic atrial fibrillation (PAF) is superior to antiarrhythmic drug therapy with regards to effectiveness and clinical outcomes. Atrial fibrillation is the most common cardiac arrhythmia, with high rates of concomitant heart failure, stroke and mortality. During an ablation procedure, a patient can be managed with intravenous sedation or General Anesthesia (GA). Within this setting, General anesthesia is associated with improved procedure time and cure rate compared to sedation.

Airway management during GA can be achieved through a laryngeal mask airway (LMA) or an endotracheal tube (ETT). The use of LMA compared to ETT has been shown in different surgical populations to decrease procedure and recovery time, improve hemodynamic stability and reduce anesthetic requirements. It has also shown to decrease airway complications, and postoperative nausea/vomiting which are important factors that affect overall patient satisfaction.

Although general anesthesia in electrophysiology procedures is associated with a higher cure rate, there have been reports of increased airway trauma.Additionally, it is believed that volatile anesthetics may be associated with increased ventricular action potential duration as well as prolonged QT interval. The increased usage of opioids during general anesthesia is also thought to interfere with electrophysiology studies by affecting vagal tone.

At Virginia Commonwealth University (VCU) Health system, Anesthesiologists have been successfully using LMA (General Anesthesia) for ablation in PAF in eligible patients for over five years. The investigators plan to perform a retrospective review of all patients who underwent catheter ablation of PAF at Virginia Commonwealth University Health System from January 2014 - December 2015. The primary endpoint evaluated will be procedure time. Other data collected will include demographics, cardiac history, type of anesthesia, amount of intra-procedure opioids, time to discharge from post anesthesia care unit (PACU), total length of hospital stay, intra-procedure hemodynamics, intra-procedure ionotrope/chronotrope/pressor requirements. and atrial fibrillation recurrence at a 3 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary ablation for paroxysmal atrial fibrillation
* Able to obtain consent in English language
* BMI <35

Exclusion Criteria:

* Patients <18 years old
* Patients undergoing ablation for arrhythmias other than paroxysmal atrial fibrillation
* American Society of Anesthesiologist physical status of 4 or greater
* Patients undergoing repeat ablation
* BMI >35
* Pregnancy
* Prisoners
* Patients unable to give their own consent
* Patients having trans esophageal echo on the same day
* Patients unable to give consent in English language
* Patients will also be excluded if the attending anesthesiologist determines that they would not be suitable candidates for intubation with either method (ETT tube or LMA mask).
* Patients with severe gastroesophageal reflux disease
* Patients with high risk of aspiration

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Prasanna, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (1.3) | 61.6 (1.8) | 63.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 27 | 27 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 38 | 46 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Procedure Time (Minutes)
Description: Will be measured as time from start of procedure to end of procedure, as recorded in minutes
Time Frame: Up to 270 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
minutes | 128.7 (4.2) | 137.8 (6.1)

2. Secondary Outcome: Fluoroscopy Time
Description: As measured and reported by electrophysiology and radiology notes, recorded in minutes
Time Frame: Up to 270 minutes
Measure: Mean (Standard Error); unit: minutes
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
minutes | 27.1 (1.7) | 28.7 (1.9)

3. Secondary Outcome: Total Anesthesia Time
Description: Total anesthesia time as measured in minutes and recorded in the anesthesia record, from anesthesia start time to anesthesia stop time
Time Frame: Up to 270 minutes
Measure: Mean (Standard Error); unit: minutes
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
minutes | 179 (4.9) | 184.7 (6.3)

4. Secondary Outcome: Time to Discharge From PACU
Description: time from arrival to PACU until discharge from anesthesia care
Time Frame: Up to 7 days
Population: Data not collected for this variable
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Total Intra-procedure Opioids
Description: Measured in mcg of Fentanyl
Time Frame: Up to 270 minutes
Measure: Mean (Standard Error); unit: mcg
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
mcg | 111.7 (6.8) | 109.2 (5.4)

6. Secondary Outcome: Anesthetic Requirements
Description: average end tidal volatile anesthetics Measured as intra operative anesthetic (MAC)
Time Frame: Up to 270 minutes
Measure: Mean (Standard Error); unit: Minimum Alveolar Concentration (MAC)
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
Minimum Alveolar Concentration (MAC) | 0.78 (0.02) | 0.76 (0.03)

7. Secondary Outcome: Anesthetic Requirements
Description: average amount of intravenous anesthetics
Time Frame: Up to 270 minutes
Population: Data not collected for this variable
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Intraoperative Hemodynamics
Description: heart rate (beats per minute)
Time Frame: Up to 270 minutes
Population: Data was not collected
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Intraoperative Hemodynamics
Description: mean arterial pressure
Time Frame: Up to 270 minutes
Population: Data was not collected
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Intraoperative Hemodynamics
Description: systolic blood pressure
Time Frame: Up to 270 minutes
Population: Data was not collected
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Intraoperative Hemodynamics
Description: diastolic blood pressure
Time Frame: Up to 270 minutes
Population: Data was not collected
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Intraprocedure Pressor/Ionotrope/Chronotrope Requirements
Description: total measured amounts of all pressors/ionotropes and chronotropes administered intraoperatively
Time Frame: Up to 270 minutes
Measure: Mean (Standard Error); unit: milligrams
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
milligrams
  total intra-procedule ephedrine | 8.8 (2.2) | 5.4 (1.6)
  total intra-procedule phenylephrine | 0.2 (0.03) | 5.5 (5.2)

13. Secondary Outcome: Electrophysiology Parameters
Description: duration of paroxysmal atrial fibrillation prior to procedure
Time Frame: Up to 270 minutes
Population: Data was not collected
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Electrophysiology Parameters
Description: size of left atrium (mm)
Time Frame: Up to 270 minutes
Population: Data was not collected
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Electrophysiology Parameters
Description: left ventricular ejection fraction
Time Frame: Up to 270 minutes
Population: Data was not collected
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Airway Trauma
Description: Any noted trauma in the anesthesia or post-procedure notes, including damage to lips/teeth, laryngospasm, need for reintubation post procedure
Time Frame: Up to 7 days
Measure: Number; unit: Incidents
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
Incidents | 0 | 0

17. Secondary Outcome: Post-procedure Nausea
Description: Measured by number of doses of antiemetics given in the post-procedure time period mg of Zofran (ondanesteron) given post-operatively
Time Frame: Up to 7 days
Measure: Mean (Standard Error); unit: Milligrams
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
Milligrams | 0.3 (0.2) | 0.9 (0.3)

18. Secondary Outcome: Post-procedure Emesis
Description: Measured by number of times patient has emesis during post-procedure time period
Time Frame: Up to 7 days
Population: Data not collected for this variable
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Atrial Fibrillation Recurrence
Description: defined as recurrence of paroxysmal atrial fibrillation recurring at any time after 6 weeks past the day of procedure. As standard of care these patients are followed up with Holter monitoring for a period of 6 months. Holter monitoring will be done for 48 hour time periods immediately post-procedure, 2 weeks, 6 weeks, 4 months and 6 months post procedure as is standard of care
Time Frame: From end of procedure to six month followup holter monitor
Measure: Number; unit: incidents
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
incidents | 2 | 2

20. Secondary Outcome: Aspiration Events
Description: aspiration events as noted in the anesthesia, PACU and post procedure notes would be documented
Time Frame: Up to 7 days
Measure: Number; unit: Events
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 50 | 50
Events | 0 | 0

21. Secondary Outcome: Patient Satisfaction
Description: patients will be given an survey by study personnel prior to discharge from the hospital; survey will be conducted in person by study personnel
Time Frame: Up to six months
Population: Not all participant provided survey data
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 43 | 44
Participants
  Very satisfied | 34 | 36
  Satisfied | 9 | 6
  Very dissatisfied | 0 | 2

22. Secondary Outcome: Cost Analysis
Description: an analysis of cost to patient as well as overall hospital costs will be conducted
Time Frame: Up to six months
Population: Data not collected
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | General Anesthesia With Endotracheal Tube | General Anesthesia With Laryngeal Mask Airway
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/95/NCT02896595/Prot_SAP_000.pdf